CLINICAL TRIAL: NCT02211976
Title: Comparative Efficacy and Tolerability of Bisacodyl Sugar Coated Tablets, Simeticone Chewing Tablets and the Combination of Both in the Treatment of Constipation and Bloatedness: an Open, Randomised, Parallel Group Trial
Brief Title: Efficacy and Tolerability of Bisacodyl Sugar Coated Tablets, Simeticone Chewing Tablets and Their Combination in Constipation and Bloatedness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 122.52
Record Dates: First submitted 2014-08-07; First posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Bisacodyl; Simethicone

ARMS (3):
- Bisacodyl (Experimental)
  Interventions: Drug: Bisacodyl
- Simeticone (Experimental)
  Interventions: Drug: Simeticone
- Bisacodyl and simeticone (Experimental)
  Interventions: Drug: Bisacodyl; Drug: Simeticone

INTERVENTIONS:
Drug: Bisacodyl
  Arms: Bisacodyl; Bisacodyl and simeticone
Drug: Simeticone
  Arms: Bisacodyl and simeticone; Simeticone

SUMMARY:
Pilot study to evaluate the efficacy and tolerability of the combined treatment of bisacodyl and simeticone compared with the efficacy and tolerability of the single products in patients suffering from constipation and bloatedness

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of constipation, defined as acute and habitual constipation; concomitantly patient must have complaint of bloated feeling
* Patient was to be 18 years of age or older
* Females who were of child bearing potential must have a negative pre-study urine pregnancy test and must be using oral or barrier contraceptive methods throughout the study. If oral contraceptives were used, the patient must be using them for at least 3 months prior to enrolment into the study
* Patient must be willing to maintain a diary throughout the study
* Patient must be otherwise in good health
* Patient must sign an informed consent form which has been prepared in accordance with the Declaration of Helsinki

Exclusion Criteria:

* Patient had drug-induced constipation resulting from drugs such as opioids, dopaminergics, antacids, anticholinergics or diuretics
* Patient had a history of organic diseases of the colon such as tumors, stricture, and acute or chronic inflammatory diseases, ileus, acute surgical abdominal conditions such as acute appendicitis, or organic diseases of the rectum and anus such as fissures, fistulas, perianal abscesses, and eczema of the perianal skin
* Patient exhibited evidence of active gastrointestinal disease
* Patient was diagnosed as having intestinal obstruction, had any undiagnosed abdominal symptoms, or was in severe dehydration
* Patient had a history of major gastrointestinal surgery
* Patient had a history of hypersensitivity to substances of the triarylmethane class
* Patient had a history of hypersensitivity to substances of the class of parahydroxybenzoic esters (para group allergy)
* Patient had a history of drug or alcohol abuse
* Patient had received bisacodyl for the treatment of another indication or in a previous study within the last 7 days before enrolment.
* Patient had ingested any drug in the past week before enrolment that in the opinion of the investigator would have an effect on gastrointestinal motility (e.g. anti-cholinergic medications, opioids, smooth muscle relaxants or antacids)
* Patient required the use of a drug, other than study drug, or dietary supplement to relieve the symptoms of constipation at any time during the baseline or treatment phases of this study
* Patient was currently taking any form of tetracycline antibiotics
* Patient was a nursing mother
* Patient had received any investigational drug within the previous 4 weeks prior to enrolment
* Patient had any condition that would interfere with the completion of this study, or that would decrease the likelihood of obtaining valid results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-10; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Change in bloatedness score on a 4-point-scale | baseline, 1 hour after drug administration

SECONDARY OUTCOMES:
Change in bloatedness score on a 4-point-scale | baseline, 2 hours, 3 hours, at time of defecation
Time to defecation | up to 7 days
Number of withdrawals due to inadequate efficiency | up to 7 days
Patient's global assessment of efficacy on a 4-point-scale | up to 7 days
Number of patients with adverse events | up to 7 days
Number of patients with abnormal laboratory findings | up to 7 days
Number of withdrawals due to safety reasons | up to 7 days
Patient's assessment of overall tolerability on a 4-point-scale | up to 7 days
Investigator's assessment of overall tolerability on a 4-point-scale | up to 7 days
Number of patients with clinically significant changes in vital signs | up to 7 days